CLINICAL TRIAL: NCT03855280
Title: Evaluation of a Recombinant Factor IX Product, APVO101, in Previously-Treated Pediatric Patients With Hemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medexus Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APVO101-903
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — IB1001

STUDY DESIGN:
Intervention Model Description: Phase 3/4, single arm, open-label study with three defined phases:
  * PK Phase: Initial PK evaluation - single dose of APVO101
  * Treatment Phase: APVO101 prophylaxis treatment for 50 ED
  * Continuation Phase: After completion of the Treatment Phase, subjects may continue APVO101 prophylaxis treatment (for an additional ≥ 50 ED)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APVO101 (Experimental): APVO101: 35 - 75 IU/kg; twice weekly
  Interventions: Drug: APVO101

INTERVENTIONS:
Drug: APVO101 — Subjects will receive a single IV dose of APVO101 twice weekly or at a frequency of infusions as determined appropriate by the investigator for the particular study subject for a total of 50 ED. The starting prophylaxis dose will be based on APVO101 recovery from PK Phase assessments (only pre-infusion and 15-30 minute post-infusion samples).
  Other Names: IB1001; Recombinant factor IX; IXINITY

SUMMARY:
Phase 3/4, single arm, open-label study to evaluate PK, safety, and efficacy of APVO101 prophylaxis in severe or moderately severe hemophilia B subjects < 12 years of age.

DETAILED DESCRIPTION:
Study APVO101-903 is a Phase 3/4, single arm, open-label clinical trial. The purpose of the study is to evaluate pharmacokinetics (PK), safety, and efficacy of APVO101 prophylaxis in severe or moderately severe hemophilia B subjects < 12 years of age. The study is designed to gather information in two age groups of previously treated (with a minimum of 50 previous ED to factor IX replacement therapy) pediatric patients, specifically those < 6 years of age and 6 to <12 years of age.

Study APVO101-903 consists of three distinct phases:

* PK Phase - PK evaluation will consist of administration of a single 75 ± 5 IU/kg dose, followed by factor IX activity and safety assessments up to 50 hours post-infusion.
* Treatment Phase - subjects will receive APVO101 prophylaxis (starting prophylaxis dose to be determined based on APVO101 recovery; ideally within the recommended dose range: 35 - 75 IU/kg; twice weekly) for 50 ED (approximately 6 months).
* Continuation Phase - subjects may continue to receive APVO101 prophylaxis (recommended dose range: 35 - 75 IU/kg; twice weekly) for an additional ≥ 50 ED.

ELIGIBILITY:
Inclusion Criteria:

1. Age: < 11.5 years of age at the time of the first dose and < 12 years throughout the Treatment Phase of the study (for at least 50 ED).
2. Informed consent: subject's parent or legal guardian written Institutional Review Board (IRB)/Ethics Committee (EC)-approved informed consent. An assent form (IRB/EC-approved) will be obtained, when required by local regulations/guidelines.
3. Willingness and ability to make the required study visits, and follow instructions while enrolled in the study (for at least 50 ED; approximately 6 months).
4. Documented severe or moderately severe hemophilia B diagnosis (factor IX activity ≤ 2 IU/dL); in addition, severity may be indicated by the occurrence of one or more joint bleeding episode(s) at any point in the child's medical history requiring infusion(s) to replace factor IX.
5. Subjects must be on prophylaxis or switch to a prophylaxis regimen for the duration of the study.
6. Previously treated patients with a minimum of 50 ED (as documented and determined by the investigator) to a preparation/blood components containing factor IX.
7. Willingness to adhere to the 4-day washout period of any factor IX replacement therapy prior to PK evaluation. In case of previous exposure to a factor IX product with a prolonged half-life, a washout period of 3 half-lives is required in order to achieve steady state factor IX level prior to exposure to APVO101.
8. Immunocompetent (CD4 count > 400/mm3) and not receiving immune modulating or chemotherapeutic agents.
9. Platelet count at least 150,000/mm3.
10. Liver function: alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2 times the upper limit of the normal range.
11. Total bilirubin ≤ 1.5 times the upper limit of the normal range.
12. Renal function: serum creatinine ≤ 1.25 times the upper limit of the normal range.
13. Hemoglobin ≥ 7 g/dL.

Exclusion Criteria:

1. History of factor IX inhibitor ≥ 0.6 Bethesda Units (BU); confirmed by the screening result.
2. Existence of another coagulation disorder.
3. Evidence of thrombotic disease, fibrinolysis, or disseminated intravascular coagulation (DIC).
4. Use of an investigational drug within 30 days prior to study entry.
5. Previous use of APVO101.
6. Use of medications that could impact hemostasis, such as aspirin.
7. Known hypersensitivity to the active substance or to any of the excipients in the investigational products.
8. Known allergic reaction to hamster proteins.
9. History of poor compliance, geographic isolation, unreliable transportation, a serious medical or social condition, or any other circumstance that, in the opinion of the investigator, would interfere with participation or compliance with the study protocol.
10. History of adverse reaction to either plasma-derived factor IX or recombinant factor IX that interfered with the subject's ability to treat bleeding episodes with a factor IX product.
11. History of any medical condition that would impact the efficacy evaluation and/or safety evaluation of the study product.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Mohamed, Study Chair — Medexus Pharma, Inc.
Locations (11):
- Brazil (3):
  - Centro Estadual de Hemopterapia e Hematologia do Espirito Santo, Vitória, Espírito Santo
  - Universidade Estadual de Campinas - Centro de Hematologia e Hemoterapia, Campinas
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto
- JSC K Eristavi National Center for Experimental and Clinical Surgery, Tbilisi, Georgia
- PMSI Institute of Mother and Child, Chisinau, Moldova
- South Africa (2):
  - Worthwhile Clinical Trials, Lakeview Hospital, Benoni, Gauteng
  - Haemophilia Comprehensive Care Centre, Johannesburg
- Turkey (Türkiye) (2):
  - Cukurova University School of Medicine, Adana
  - Ege University School ofMedicine, Izmir
- Ukraine (2):
  - National Specialized Children's Hospital OKHMATDYT, Kyiv
  - State Institute: Institute of Blood Pathology and Transfusion Medicine of the National Academy of Medical Sciences of Ukraine, Lviv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pediatric patients (less than 11.5 years of age at first dose) with severe to moderately severe hemophilia B.
  Participants had a minimum of 50 exposure days of factor IX (FIX) replacement therapy prior to enrollment.
Groups:
- APVO101 Prophylaxis - Safety Population: Following a four day washout period or three half-lives washout of a factor IX product with a prolonged half-life, all study participants entered the PK Phase.
  * PK Phase - PK evaluation consisted of administration of a single 75 (±5) IU/kg dose, followed by factor IX activity and safety assessments up to 50 hours post-infusion.
  * Treatment Phase - after completion of the PK Phase, participants (safety population) received APVO101 prophylaxis (starting prophylaxis dose was to be determined based on APVO101 recovery; ideally within the recommended dose range: 35 to 75 IU/kg, twice weekly or at a frequency determined as appropriate by the Investigator) for 50 exposure days (approximately 6 months).
  * Continuation Phase - participants could continue APVO101 prophylaxis (recommended dose range: 35 to 75 IU/kg, twice weekly) for an additional 50 or more exposure days (approximately 6 months).
Period: PK Phase
Arm/Group | APVO101 Prophylaxis - Safety Population
Started | 21 (Age group < 6 years of age (N=10) Age group 6 to < 12 years of age (N=11))
PK Phase | 21
Completed | 21 (Age group < 6 years of age (N=10) Age group 6 to < 12 years of age (N=11))
Not Completed | 0
Period: Treatment Phase
Arm/Group | APVO101 Prophylaxis - Safety Population
Started | 21
Completed (21 subjects entered the Treatment Phase; 19 subjects completed the study (i.e., completion of PK assessments and a minimum of 50 ED).) | 19
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Continuation Phase
Arm/Group | APVO101 Prophylaxis - Safety Population
Started | 19
Completed | 16
Not Completed | 3
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 1
Not completed — Sponsor Concluded Study | 1

BASELINE CHARACTERISTICS:
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 21
Age, Customized [Count of Participants; unit: Participants]
  Age Group: < 6 | 10
  Age Group: 6 to < 12 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 4
  Ukraine | 8
  Brazil | 3
  South Africa | 3
  Moldova | 1
  Georgia | 2
Retrospective Annualized Bleeding Rate [Mean (Standard Deviation); unit: bleeding episodes per year] — No quantifiable data were measured or analyzed. Population: There was no quantifiable retrospective data to report for this table.

OUTCOME MEASURES:

1. Primary Outcome: Annualized Bleeding Rate (ABR)
Description: The primary efficacy variable was the ABR while on prophylaxis to prevent bleeding episodes. The ABR was defined as the number of bleeding episodes per year.
Time Frame: Exposure Day 1 up to 50 exposure days (approximately 6 months)
Population: Analysis population included all participants for whom a legally acceptable representative had signed the informed consent/assent form and received at least one dose of APVO101.
Measure: Mean (Standard Deviation); unit: bleeding episodes per year
Groups:
- APVO101 - Safety Population: Following a four day washout period or three half-lives washout of a factor IX product with a prolonged half-life, all study participants entered the PK Phase.
  * PK Phase - PK evaluation consisted of administration of a single 75 (±5) IU/kg dose, followed by factor IX activity and safety assessments up to 50 hours post-infusion.
  * Treatment Phase - after completion of the PK Phase, participants (safety population) received APVO101 prophylaxis (starting prophylaxis dose was to be determined based on APVO101 recovery; ideally within the recommended dose range: 35 to 75 IU/kg, twice weekly or at a frequency determined as appropriate by the Investigator) for 50 exposure days (approximately 6 months).
  * Continuation Phase - participants could continue APVO101 prophylaxis (recommended dose range: 35 to 75 IU/kg, twice weekly) for an additional 50 or more exposure days (approximately 6 months).
Arm/Group | APVO101 - Safety Population
Number analyzed (Participants) | 21
bleeding episodes per year | 2.93 (4.59)

2. Primary Outcome: Annualized Bleeding Rate (ABR) Overall
Description: as for outcome 1
Time Frame: Exposure Day 1 through study completion (up to 2.5 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bleeding episodes per year
Arm/Group | APVO101 - Safety Population
Number analyzed (Participants) | 21
bleeding episodes per year | 2.34 (4.23)

3. Secondary Outcome: Concentration (Cmax)
Description: Maximum post-infusion plasma concentration of FIX activity was measured at the following time points post infusion: 15-30 minutes, 4-6 hours, 24-26 hours and 46-50 hours.
Time Frame: Pre-infusion to 50 hours post-infusion
Population: Analysis population included all participants for whom legally acceptable representative had signed informed consent/assent form, were in non-bleeding state, participated in single PK assessment at start of study and for whom an adequate PK profile had been obtained. "Number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | APVO101 - Safety Population
Number analyzed (Participants) | 20
IU/dL | 60.1 (12.2)

4. Secondary Outcome: Area Under the Curve (0-inf)
Description: Area under plasma concentration curve, FIX activity-time profile from time zero extrapolated to infinity. FIX activity was measured at the following time points post infusion: 15-30 minutes, 4-6 hours, 24-26 hours and 46-50 hours.
Time Frame: Pre-infusion to 50 hours post-infusion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/dL/hr
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 21
IU/dL/hr | 1170 (231)

5. Secondary Outcome: Mean Residence Time (MRT)
Description: MRT is the average time the molecules of drug reside in the body before elimination.
Time Frame: Pre-infusion to 50 hours post-infusion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 11
hours | 20 (2.53)

6. Secondary Outcome: Terminal Half-Life (t 1/2)
Description: Terminal half-life is the length of time required for the concentration of drug to decrease by one half of its starting dose in the body. FIX activity was measured at the following time points post infusion: 15-30 minutes, 4-6 hours, 24-26 hours and 46-50 hours.
Time Frame: Pre-infusion to 50 hours post-infusion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 12
hours | 16.3 (2.2)

7. Secondary Outcome: Clearance (CL)
Description: Clearance is a measure of the volume of plasma from which FIX activity is removed per unit time. Weight normalized clearance calculated as CL=Dose/AUC 0-inf. FIX activity was measured at the following time points post infusion: 15-30 minutes, 4-6 hours, 24-26 hours and 46-50 hours.
Time Frame: Pre-infusion to 50 hours post-infusion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/(kg*hr)
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 11
mL/(kg*hr) | 6.8 (1.5)

8. Secondary Outcome: Volume of Distribution at Steady-State (Vdss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of FIX would need to be uniformly distributed to produce the observed plasma concentration of FIX. Steady state volume of distribution (Vdss) is the apparent volume of distribution at steady-state. FIX activity was measured at the following time points post infusion: 15-30 minutes, 4-6 hours, 24-26 hours and 46-50 hours.
Time Frame: Pre-infusion to 50 hours post-infusion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 11
mL/kg | 134 (30.6)

9. Secondary Outcome: Incremental Recovery (IR)
Description: Incremental recovery was the increase in circulating FIX activity for every international unit (IU) of APVO101 administered per kilogram of body weight of participant. FIX activity was measured at the following time points post infusion: 15-30 minutes, 4-6 hours, 24-26 hours and 46-50 hours.
Time Frame: Pre-infusion to 50 hours post-infusion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 20
IU/dL per IU/kg | 0.790 (0.156)

10. Secondary Outcome: Subject Rating of APVO101 Efficacy - Evaluated at the Bleeding Episode Level (Treatment Phase)
Description: Subjects rated APVO101 efficacy for each bleeding episode based on a four-point scale:
  1. Excellent: a dramatic response with abrupt pain relief and clear reduction in joint or hemorrhage site size
  2. Good: pain relief or reduction in hemorrhage site size that may have required an additional infusion for resolution;
  3. Fair: probable or slight beneficial response usually requiring one of more additional infusions for resolution;
  4. Poor: no improvement or condition worsens.
Time Frame: Exposure Day 1 up to 50 exposure days (approximately 6 months)
Population: Analysis population included all participants for whom a legally acceptable representative had signed the informed consent/assent form, received at least one dose of APVO101 and who had experienced at least one bleeding episode.
Measure: Count of Units; unit: bleeding episodes
Units Other Than Participants: bleeding episodes
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 11
Number analyzed (bleeding episodes) | 24
bleeding episodes
  Excellent | 10
  Good | 5
  Fair | 0.0
  Poor | 0.0
  No infusions required to treat bleeding episode | 7
  Missing | 2

11. Secondary Outcome: Subject Rating of APVO101 Efficacy - Evaluated at the Bleeding Episode Level (Overall)
Description: as for outcome 10
Time Frame: Exposure Day 1 through study completion (up to 2.5 years)
Population: as for outcome 10
Measure: Count of Units; unit: bleeding episodes
Units Other Than Participants: bleeding episodes
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 14
Number analyzed (bleeding episodes) | 52
bleeding episodes
  Excellent | 28
  Good | 13
  Fair | 0.0
  Poor | 0.0
  No infusions required to treat bleeding episode | 9
  Missing | 2

12. Secondary Outcome: Investigator Rating of APVO101 Prophylaxis Efficacy (Treatment Phase)
Description: The investigator will indicate the overall assessment of APVO101 prophylaxis efficacy, considering the absence of bleeding episodes, site, severity and types of bleeding episodes treated, and other factors that might influence the therapeutic response.
  The investigator's efficacy assessment categories for prophylaxis will include: 'effective', 'partially effective' and 'not effective'.
Time Frame: Exposure Day 1 up to 50 exposure days (approximately 6 months)
Population: Analysis population included all participants for whom a legally acceptable representative had signed the informed consent/assent form and had received at least one dose of APVO101.
Measure: Count of Units; unit: prophylactic efficacy assessment
Units Other Than Participants: prophylactic efficacy assessment
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 21
Number analyzed (prophylactic efficacy assessment) | 81
prophylactic efficacy assessment
  Effective | 80
  Partially Effective | 1
  Not Effective | 0

13. Secondary Outcome: Investigator Rating of APVO101 Prophylaxis Efficacy (Overall)
Description: as for outcome 12
Time Frame: Exposure Day 1 through study completion (up to 2.5 years)
Population: as for outcome 12
Measure: Count of Units; unit: prophylactic efficacy assessment
Units Other Than Participants: prophylactic efficacy assessment
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 21
Number analyzed (prophylactic efficacy assessment) | 170
prophylactic efficacy assessment
  Effective | 167
  Partially Effective | 3
  Not Effective | 0

14. Secondary Outcome: Investigator Rating of APVO101 Efficacy for Control and Management of Bleeding Episodes (Treatment Phase)
Description: Of the bleeding episodes requiring treatment, the investigator considered the site, severity and type of the bleeding episode while evaluating efficacy for control and management of the bleeding episode.
  The investigator's efficacy assessment categories control of bleeding episodes included: 'effective', 'partially effective' and 'not effective'.
Time Frame: Exposure Day 1 up to 50 exposure days (approximately 6 months)
Population: as for outcome 10
Measure: Count of Units; unit: efficacy for control of bleeding episode
Units Other Than Participants: efficacy for control of bleeding episode
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 11
Number analyzed (efficacy for control of bleeding episode) | 16
efficacy for control of bleeding episode
  Effective | 16
  Partially effective | 0
  Not effective | 0

15. Secondary Outcome: Investigator Rating of APVO101 Efficacy for Control and Management of Bleeding Episodes (Overall)
Description: as for outcome 14
Time Frame: Exposure Day 1 through study completion (up to 2.5 years)
Population: as for outcome 10
Measure: Count of Units; unit: efficacy for control of bleeding episode
Units Other Than Participants: efficacy for control of bleeding episode
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 14
Number analyzed (efficacy for control of bleeding episode) | 35
efficacy for control of bleeding episode
  Effective | 35
  Partially effective | 0
  Not effective | 0

16. Other Pre Specified Outcome: Spontaneous Annualized Bleeding Rate (Treatment Phase)
Description: Includes annualized bleeding rate for spontaneous bleeding (i.e. bleeds that occur without obvious cause).
Time Frame: Exposure Day 1 up to 50 exposure days (approximately 6 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: spontaneous bleeding episodes
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 21
spontaneous bleeding episodes | 0.81 (1.93)

17. Other Pre Specified Outcome: Spontaneous Annualized Bleeding Rate (Overall)
Description: Includes annualized bleeding rate for spontaneous bleeding (i.e. bleeds that occur without obvious cause).
Time Frame: Exposure Day 1 through study completion (up to 2.5 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: spontaneous bleeding episodes
Arm/Group | APVO101 Prophylaxis - Safety Population
Number analyzed (Participants) | 21
spontaneous bleeding episodes | 0.63 (1.26)

18. Other Pre Specified Outcome: Occurrence of Inhibitory Factor IX Antibodies (Overall)
Description: Incidence of APVO101 immunogenicity response (development of inhibitory, non-inhibitory factor IX binding antibodies and incidence of antibodies to Chinese hamster ovary cell proteins [CHOP])
Time Frame: Exposure Day 1 through study completion (up to 2.5 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | APVO101 - Safety Population
Number analyzed (Participants) | 21
Participants | 0

19. Other Pre Specified Outcome: Occurrence of Non-Inhibitory Factor IX Antibodies (Overall)
Description: as for outcome 18
Time Frame: Exposure Day 1 through study completion (up to 2.5 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | APVO101 - Safety Population
Number analyzed (Participants) | 21
Participants | 3

20. Other Pre Specified Outcome: Occurrence of Anti-CHOP Antibodies (Overall)
Description: as for outcome 18
Time Frame: Exposure Day 1 through study completion (up to 2.5 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | APVO101 - Safety Population
Number analyzed (Participants) | 21
Participants | 3

21. Other Pre Specified Outcome: Thrombogenicity Assessment - D-Dimer
Description: This study included testing of thrombogenic markers at the PK stage to evaluate for thrombotic risk.
Time Frame: Day 1 (pre-dose), 15-30 minutes, 4-6 hours and 24-26 hours post-infusion
Population: To accommodate blood volume limitations for participants less than 17 kg, no thrombogenicity assessments were performed during the PK Phase. Participants weighing 17 kg to 19 kg, the 4 to 6 hour post-infusion timepoint was not collected.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Actual Value: Prespecified collection timepoint value
- Change From Baseline: Change from Baseline in values during the prespecified collection timepoints
Arm/Group | Actual Value | Change From Baseline
Number analyzed (Participants) | 13 | 13
mg/L
  Day 1, pre-infusion: number analyzed (Participants) | 13 | 0
  Day 1, pre-infusion | 0.432 (0.2320) |
  15 to 30 minutes post-infusion | 0.422 (0.1999) | 0.006 (0.1071)
  4 to 6 hours post-infusion: number analyzed (Participants) | 13 | 11
  4 to 6 hours post-infusion | 0.452 (0.2955) | 0.045 (0.2051)
  24 to 26 hours post-infusion | 0.578 (0.2766) | 0.114 (0.2586)

22. Other Pre Specified Outcome: Thrombogenicity Assessment - Thrombin/Antithrombin (TAT) Complex
Description: This study included testing of thrombogenic markers at the PK stage to evaluate for thrombotic risk.
Time Frame: Day 1 (pre-dose), 15-30 minutes, 4-6 hours and 24-26 hours post-infusion
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Actual Value | Change From Baseline
Number analyzed (Participants) | 13 | 13
ug/L
  Day 1, pre-infusion: number analyzed (Participants) | 13 | 0
  Day 1, pre-infusion | 5.92 (2.579) |
  15 to 30 minutes post-infusion | 17.92 (22.971) | 12.71 (24.252)
  4 to 6 hours post-infusion: number analyzed (Participants) | 13 | 11
  4 to 6 hours post-infusion | 12.17 (15.986) | 6.63 (17.399)
  24 to 26 hours post-infusion | 12.45 (16.459) | 6.78 (17.081)

23. Other Pre Specified Outcome: Thrombogenicity Assessment - Prothrombin Fragment 1+2
Description: This study included testing of thrombogenic markers at the PK stage to evaluate for thrombotic risk.
Time Frame: Day 1 (pre-dose), 15-30 minutes, 4-6 hours and 24-26 hours post-infusion
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Actual Value | Change From Baseline
Number analyzed (Participants) | 13 | 13
pmol/L
  Day 1, pre-infusion: number analyzed (Participants) | 13 | 0
  Day 1, pre-infusion | 99.9 (41.59) |
  15 to 30 minutes post-infusion | 318.0 (433.64) | 218.1 (439.48)
  4 to 6 hours post-infusion: number analyzed (Participants) | 13 | 11
  4 to 6 hours post-infusion | 238.6 (330.63) | 139.5 (303.66)
  24 to 26 hours post-infusion | 223.0 (246.46) | 123.1 (251.48)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored after the first dose of APVO101 through study completion (up to 2.5 years) with a minimum follow-up period of 30 days.
Description: Collection method: All adverse events were reported by investigators assessments and subjects and/or their parent or legal guardian. Any clinically significant changes (as determined by the investigator) in laboratory test results, vital signs or physical exam were captured as adverse events. Additionally, subjects and/or their parent or legal guardian recorded AEs in the subject diary and the information was reviewed by the investigator during each scheduled visit.
Groups:
- APVO101 Prophylaxis - Safety Population: All subjects in the Safety Population received study treatment.
Arm/Group | APVO101 Prophylaxis - Safety Population
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APVO101 Prophylaxis - Safety Population (N=21)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) — The TEAE was considered by the investigator and sponsor to be unrelated to APVO101.
Hematuria (Renal and urinary disorders) | 1 (1) — The TEAE was considered by the investigator and sponsor to be unrelated to APVO101.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APVO101 Prophylaxis - Safety Population (N=21)
Bronchitis (Infections and infestations) | 12 (31)
Influenza (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (7)
Respiratory tract infection (Infections and infestations) | 2 (4)
Respiratory tract infection viral (Infections and infestations) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT03855280/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT03855280/SAP_001.pdf